CLINICAL TRIAL: NCT03515616
Title: Evaluation of Role of TP US in Progress of Labour by PC Angle & OS Angle
Brief Title: Evaluation of Labour Progress by PC Angle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, National Research Centre, Egypt
Other Study IDs: labour assesment by US
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Labour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TP us in labour — TP US will be made to pregnant lady in first stage of labour with OS and PC angel measurements

SUMMARY:
- Ultrasound during first stage of labour has a very important role in prediction of mode of delivery

DETAILED DESCRIPTION:
-Operative delivery and cs delivery are increasing nowadays so US during labour is vital to predict these interventions

ELIGIBILITY:
Inclusion Criteria:

* primigravida
* pregnant full term
* no medical disorders

Exclusion Criteria:

* multigravida
* any medical disorders
* preterm labour

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant ladies ful term
Study Population: - primigravida who is pregnant full term with no medical disorders
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-05-10 (Estimated); Study Completion 2019-06-14 (Estimated)

PRIMARY OUTCOMES:
the number of participants who will deliver by NVD without instrumental intervention | within 36 hours
  the number of pregnant ladies in first stage of labour who will deliver by NVD and who will have normal progress or prolonged progress of labour

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, M.s.c, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (2):
- Egypt (2):
  - Kasralainy Hospital, Cairo
  - Algazeerah, Giza

IPD SHARING:
Plan to Share IPD: No
data which will be obtained from this study will be published